CLINICAL TRIAL: NCT00452387
Title: Mitoxantrone, Prednisone Plus Sorafenib in Taxane-Refractory Metastatic Hormone Refractory Prostate Cancer (HRPC)
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Early stopping rule
Sponsor: Accelerated Community Oncology Research Network (Other)
Collaborators: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ACORN AVAHRPC0607
Record Dates: First submitted 2007-03-26; First posted 2007-03-27 (Estimated); Results first posted 2010-05-26 (Estimated); Last update posted 2011-09-16 (Estimated); Status verified 2011-09

CONDITIONS: Metastatic Prostate Cancer
Keywords: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Mitoxantrone; Prednisone; Sorafenib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Mitoxantrone — Once six patients are accrued at dose level 1, the maximum tolerated dose (MTD) will be assessed by following them through one cycle of treatment. If 2/6 patients experience dose limiting toxicity (DLT) at the 400 mg twice a day (bid) level then the MTD will be defined as 400 mg daily (QD). Additional patients will be enrolled at the MTD for the phase II portion.
  Dose Level -2, Mitoxantrone 9mg/m2
  Dose Level -1 Mitoxantrone 12mg/m2
  Dose Level 1 Mitoxantrone 12mg/m2
  Other Names: Novantrone
Drug: Prednisone — Once six patients are accrued at dose level 1, the maximum tolerated dose (MTD) will be assessed by following them through one cycle of treatment. If 2/6 patients experience dose limiting toxicity (DLT) at the 400 mg twice a day (bid) level then the MTD will be defined as 400 mg daily (QD). Additional patients will be enrolled at the MTD for the phase II portion.
  Dose Level -2, Prednisone 5mg bid
  Dose Level -1 Prednisone 5mg bid
  Dose Level 1 Prednisone 5mg bid
  Other Names: Deltasone
Drug: Sorafenib — Once six patients are accrued at dose level 1, the maximum tolerated dose (MTD) will be assessed by following them through one cycle of treatment. If 2/6 patients experience dose limiting toxicity (DLT) at the 400 mg twice a day (bid) level then the MTD will be defined as 400 mg daily (QD). Additional patients will be enrolled at the MTD for the phase II portion.
  Dose Level -2, Sorafenib 400 mg QD
  Dose Level -1 Sorafenib 400 mg QD
  Dose Level 1 Sorafenib 400 mg bid
  Other Names: Nexavar

SUMMARY:
The purpose of this research study is to determine if the combination of mitoxantrone, prednisone and sorafenib will improve the time to progression of advanced stage metastatic hormone-refractory prostate cancer.

DETAILED DESCRIPTION:
The primary objective of this study is to test the hypothesis that the combination of Mitoxantrone, Prednisone and Sorafenib in taxane-refractory patients with metastatic hormone refractory prostate cancer (mHRPC) will result in an improvement of the median time to progression (TTP). Since the median (i.e 50% of patients) TTP for Mitoxantrone/Prednisone is 3 months, our hypothesis is that 70% will have not progressed at 3 months with this investigational combination. Progression will be assessed by radiologic imaging criteria.

The early stopping point is 21 subjects. If 10 or fewer subjects with tumor favorable response are observed when 21 subjects are accrued then the null hypothesis is accepted and the trial is terminated. If 16 or more subjects with tumor favorable response are observed when 21 subjects are accrued then the alternative hypothesis is accepted and the trial is terminated. The probability of early stopping under the null is 0.51, and under the alternative is 0.39. If the trial progresses until 42 subjects are evaluated and 24 or more subjects with favorable response are observed then the null hypothesis is rejected. This design minimizes the average sample number under the null, which is 31.2.

ELIGIBILITY:
Inclusion Criteria:

* Voluntary written informed consent
* Histopathologic diagnosis of prostatic adenocarcinoma with evidence of progression despite adequate castration (testosterone < 50 ng/dL)
* Progressive disease after taxane-based chemotherapy (docetaxel or paclitaxel, single agent or combination regimens, weekly or every 21 day schedules)
* Patients who discontinued taxane- based chemotherapy because of toxicity will be eligible as long as there is evidence of progressive disease
* Minimum of 4 weeks period from last chemotherapy infusion to registration (this does not apply to steroid use which is permitted). Estramustine needs to be discontinued at least 6 weeks prior to first day of treatment on protocol
* A minimum of 4 weeks off bicalutamide, nilutamide, megestrol acetate ketoconazole, diethylstilbestrol (DES). Minimum of 2 weeks off flutamide
* Reductase inhibitors will be allowed if initiated at least 2 months prior to registration
* No concurrent investigational therapy
* Complementary and Alternative Medicine (CAM) products will be permitted as long as patients have been receiving them for at least 2 months. Initiation of new CAM products while on protocol will be discouraged.
* Ongoing androgen deprivation therapy (orchiectomy, gonadotropin-releasing hormone (GnRH) agonist or antagonist)
* Adequate bone marrow, liver and renal function as assessed by the following:

  * Hemoglobin ≥ 9.0 g/dl
  * Absolute neutrophil count (ANC) ≥ 1,500/mm3
  * Platelet count ≥ 100,000/mm3
  * Total bilirubin ≤ 1.5 times upper limit of normal (ULN)
  * ALT and AST ≤ 2.5 times the ULN ( ≤ 5 x ULN for patients with liver involvement)
  * Creatinine ≤ 1.5 times the ULN
* International normalized ratio (INR) < 1.5 or a Prothrombin (PT)/Partial thromboplastin time (PTT) within normal limits. Patients receiving anti-coagulation treatment with an agent such as warfarin or heparin may be allowed to participate. For patients on warfarin, the INR should be measured prior to initiation of sorafenib and monitored at least weekly, or as defined by the local standard of care, until INR is stable.
* ECOG performance status ≤ 2
* Baseline left ventricular ejection fraction (LVEF) ≥ 50%
* Life expectancy ≥ 3 months
* Patients must agree to use adequate contraception prior to study entry, during the study and for at least three months after the last administration of sorafenib

Exclusion Criteria:

* More than one line of prior cytotoxic chemotherapy in the metastatic setting, previous adjuvant chemotherapy will be allowed
* No active malignancy other than prostate cancer (except non-melanoma skin cancer) within 5 years of enrollment
* Known brain metastases
* Cardiac disease: Congestive heart failure > class II New York Heart Association (NYHA). Patients must not have unstable angina or new onset angina (began within the last 3 months) or myocardial infarction within the past 6 months
* Cardiac ventricular arrhythmias requiring anti-arrhythmic therapy
* Uncontrolled hypertension
* Active clinically serious infection > Common Terminology Criteria for Adverse Events (CTCAE) Grade 2
* Thrombolic or embolic events such as a cerebrovascular accident including transient ischemic attacks within the past 6 months
* Pulmonary hemorrhage/bleeding event ≥ CTCAE Grade 2 within 4 weeks of first dose of study drug
* Any other hemorrhage/bleeding event ≥ CTCAE Grade 3 within 4 weeks of first dose of study drug
* Poorly controlled hyperglycemia
* Treatment with radiotherapy within 4 weeks or treatment with radiopharmaceuticals within past 8 weeks
* Patient has received other investigational drugs within 14 days before enrollment
* Serious medical or psychiatric illness likely to interfere with participation in this clinical study
* Serious non-healing wound or ulcer
* Evidence or history of bleeding diathesis or coagulopathy
* Use of St. John's Wort or rifampin
* Known or suspected allergy to sorafenib or any agent given in the course of this trial
* Any condition that impairs patient's ability to swallow whole pills
* Any malabsorption problem

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2007-05; Primary Completion 2008-07 (Actual); Study Completion 2009-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Vasily Assikis, MD, Principal Investigator — Peachtree Hematology Oncology Consultants
Locations (10):
- United States (10):
  - Wilshire Oncology Medical Group, Inc., La Verne, California
  - Peachtree Hematology Oncology Consultants, Atlanta, Georgia
  - Central Georgia Cancer Care, Macon, Georgia
  - Northwest Georgia Oncology Centers, Marietta, Georgia
  - Hematology Oncology Centers of the Northern Rockies, PC, Billings, Montana
  - Mid-Ohio Oncology/Hematology, Inc., Columbus, Ohio
  - Lancaster Cancer Center, Lancaster, Pennsylvania
  - Pennsylvania Oncology Hematmology Associates, Philadelphia, Pennsylvania
  - The West Clinic, Memphis, Tennessee
  - Cancer Specialists of Tidewater, Chesapeake, Virginia

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 10 community oncology research sites across the US within the ACORN network participated in this study. Enrollment started in May 2007 and was closed in July 2008 after the interim analysis was completed.
Pre-assignment Details: Informed consent was obtained from all subjects. All subjects underwent a screening period that could last up to 4 weeks during which pre-study assessments were completed.
Groups:
- Treatment Group: Mitoxantrone, Prednisone, Plus Sorafenib: The treatment plan for all subjects was mitoxantrone 12 mg/m2 IV every 21 days; sorafenib 400 mg po bid daily; and prednisone 5 mg po bid daily.
Period: Overall Study
Arm/Group | Treatment Group: Mitoxantrone, Prednisone, Plus Sorafenib
Started | 22
Completed | 22
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Treatment Group: Mitoxantrone, Prednisone, Plus Sorafenib
Number analyzed (Participants) | 22
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 8
  >=65 years | 14
Age Continuous [Mean (Standard Deviation); unit: years] | 67 (9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 22
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 20
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 22

OUTCOME MEASURES:

1. Primary Outcome: Median Time to Progression (TTP) by Imaging
Description: Time to progression is defined as the time from treatment start until objective tumor progression. The median time to progression is the parameter used to describe TTP.
Time Frame: Radiologic imaging was repeated after every 4 cycles (approximately every 12 weeks) during study treatment.
Population: Survival analysis was performed for 22 patients. However, the upper 95% confidence interval for median TTP could not be calculated and so the number of patients analyzed and the upper 95% confidence interval for median TTP could not be entered into the system.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Treatment Group: Mitoxantrone, Prednisone, Plus Sorafenib
Number analyzed (Participants) | 0

2. Secondary Outcome: Correlation of Biochemical Criteria (PSA, Prostate-specific Antigen) With Objective Imaging
Description: The test of association assesses the null hypothesis that the frequency of PSA response is the same for patients with and without a favorable imaging response. PSA response required a 50% reduction of the baseline PSA result that was confirmed three weeks later. Favorable imaging response is defined as stable disease, partial response, or complete response per RECIST guidelines. The Fisher's exact test was used to test this hypothesis.
Time Frame: PSA was evaluated on day 1 of every cycle (approximately every 3 weeks) during study treatment. Radiologic imaging was repeated after every 4 cycles (approximately every 12 weeks) during study treatment.
Measure: Number; unit: Participants
Arm/Group | Imaging Response (Favorable) | Imaging Response (Unfavorable)
Number analyzed (Participants) | 9 | 13
Participants
  PSA response (> 50% reduction) | 3 | 0
  PSA response (< or = 50% reduction) | 6 | 13
Statistical Analysis 1: Comparison: Imaging Response (Favorable) vs Imaging Response (Unfavorable); The test of association of PSA and imaging response tests the null hypothesis that the proportion of cases exhibiting PSA response is the same for patients with and without a favorable imaging response. A 2x2 table was constructed based on the number of the patients in imaging response (favorable and unfavorable) and PSA response (>50% reduction and <=50% reduction). The Fisher's exact test was used to test this hypothesis; Test type: Superiority or Other; p = 0.55, Fisher Exact

3. Secondary Outcome: Quality of Life (QoL)
Description: The subject answers questions from the following 6 categories: general physical symptoms, treatment side effects, distress, despair, impaired performance, and impaired ambulation. Each question has a scale from 0 through 10, where 0 is not a problem and 10 is as bad as possible. The scores for the 6 categories are combined and normalized, and used to describe overall quality of life. Because normalized scores are created using a look-up index, there is no clearly defined maximum value. In practice, the maximum value for the combined scale is 73.5.
Time Frame: The Patient Care Monitor questionnaire was administered on day 1 of every cycle (approximately every 3 weeks) during study treatment.
Measure: Mean (Full Range); unit: units on a scale
Arm/Group | Treatment Group: Mitoxantrone, Prednisone, Plus Sorafenib
Number analyzed (Participants) | 22
units on a scale
  Baseline | 50.21 [32.95 to 60.27]
  Cycle 1 | 49.71 [30.03 to 59.36]
  Cycle 2 | 51.06 [40.11 to 60.76]
  Cycle 3 | 51.20 [34.63 to 60.08]
  Cycle 4 | 51.66 [44.31 to 57.50]
  Cycle 5 | 51.22 [42.50 to 59.36]
  Cycle 6 | 49.73 [38.59 to 55.61]
  Cycle 7 | 49.50 [38.16 to 59.36]
  Cycle 8 | 48.20 [35.91 to 59.18]
  Cycle 9 | 54.34 [52.69 to 56.01]
  Cycle 10 | 55.88 [51.38 to 59.01]
  Cycle 11 | 54.95 [54.95 to 54.95]
  Cycle 12 | 54.02 [51.47 to 56.55]
  Cycle 13 | 54.65 [54.65 to 54.65]
  End of Study (at treatment discontinuation) | 45.13 [40.20 to 53.72]

4. Secondary Outcome: Median Overall Survival (OS)
Description: Overall survival is defined as the time from treatment start until death from any cause. The median overall survival time is used to measure OS.
Time Frame: Overall survival was measured from day 1 of treatment until the end of treatment and then every 3 months thereafter until death.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Treatment Group: Mitoxantrone, Prednisone, Plus Sorafenib
Number analyzed (Participants) | 22
Months | 12.32 [7.82 to 22.50]

ADVERSE EVENTS:
Time Frame: Adverse events were collected beginning on day 1 of study treatment until one month after the end of study treatment.
Description: Systematic Assessment - subjects were assessed for adverse events on day 1 of each cycle by either the research coordiantor, treating physician, or other appropriate sub-investigator.
Arm/Group | Treatment Group: Mitoxantrone, Prednisone, Plus Sorafenib
Serious Adverse Events (participants affected / at risk) | 10/22
Other Adverse Events (participants affected / at risk) | 20/22
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment Group: Mitoxantrone, Prednisone, Plus Sorafenib (N=22)
Neutropenia (Blood and lymphatic system disorders) | 1 (1)
Acute gastritis (Gastrointestinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1)
Pain - abdominal (Gastrointestinal disorders) | 2 (2)
Vomiting (Gastrointestinal disorders) | 1 (1)
Death (General disorders) | 1 (1)
Necrosis (General disorders) | 1 (1)
Pain - chest (General disorders) | 1 (1)
Acute osteomylitis (Infections and infestations) | 1 (1)
Esophageal candidiasis (Infections and infestations) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 1 (1)
Osteonecrosis of mandible (Musculoskeletal and connective tissue disorders) | 1 (1)
Pain - hip (Musculoskeletal and connective tissue disorders) | 1 (1)
Pain - jaw (Musculoskeletal and connective tissue disorders) | 1 (1)
Pain - shoulder (Musculoskeletal and connective tissue disorders) | 1 (2)
Lower extremities paraparesis (Nervous system disorders) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Hand and foot syndrome (Skin and subcutaneous tissue disorders) | 1 (1)
Rash/desquamation (Skin and subcutaneous tissue disorders) | 1 (1)
Deep vein thrombosis of lower extremity (Vascular disorders) | 1 (1)
Dysphagia (Gastrointestinal disorders) | 1 (1)
Metastatic small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment Group: Mitoxantrone, Prednisone, Plus Sorafenib (N=22)
Anemia (Blood and lymphatic system disorders) | 3 (5)
Leukopenia (Blood and lymphatic system disorders) | 1 (2)
Neutropenia (Blood and lymphatic system disorders) | 5 (5)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (2)
Blurred vision (Eye disorders) | 1 (1)
Eye floaters (Eye disorders) | 1 (1)
Watery eyes (Eye disorders) | 1 (1)
Anal buccal tenderness (Gastrointestinal disorders) | 1 (1)
Anorexia (Metabolism and nutrition disorders) | 6 (6)
Bloating (Gastrointestinal disorders) | 1 (1)
Change in taste of food (Gastrointestinal disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 8 (10)
Dry heaves (Gastrointestinal disorders) | 1 (1)
Dysphagia (Gastrointestinal disorders) | 1 (1)
Flatulence (Gastrointestinal disorders) | 1 (1)
Gastrointestinal - abdomen NOS (intermittent) (Gastrointestinal disorders) | 1 (1)
Heartburn (Gastrointestinal disorders) | 2 (2)
Hemoccult positive stools (Gastrointestinal disorders) | 1 (1)
Melanotic stools (Gastrointestinal disorders) | 1 (1)
Mouth sores (Gastrointestinal disorders) | 2 (2)
Nausea (Gastrointestinal disorders) | 9 (12)
Pain - abdomen (Gastrointestinal disorders) | 1 (1)
Pain - esophagus (Gastrointestinal disorders) | 1 (2)
Peridontal disease (Gastrointestinal disorders) | 1 (1)
Sore mouth (Gastrointestinal disorders) | 1 (1)
Stomatitis (Gastrointestinal disorders) | 2 (2)
Vomiting (Gastrointestinal disorders) | 4 (7)
Ankle edema (General disorders) | 1 (1)
Bilateral lower extremity edema (General disorders) | 1 (1)
Fatigue (General disorders) | 13 (14)
Flu-like symptoms (General disorders) | 2 (2)
Mucositis (General disorders) | 8 (8)
Pain - chest (General disorders) | 3 (3)
Rigors without temperature (General disorders) | 1 (1)
Weakness (General disorders) | 2 (2)
Bronchitis (Infections and infestations) | 1 (1)
Diverticulitis (Infections and infestations) | 1 (1)
Herpes zoster (Infections and infestations) | 1 (1)
Positive blood cultures (Infections and infestations) | 1 (1)
Shingles (Infections and infestations) | 1 (1)
Upper respiratory infection (Infections and infestations) | 1 (1)
Urinary tract infection (Infections and infestations) | 2 (2)
T12 compression fracture (Injury, poisoning and procedural complications) | 1 (1)
Cardiac catheter (Investigations) | 1 (1)
Decreased ejection fraction (Investigations) | 1 (1)
Elevated ALT (Investigations) | 1 (1)
Elevated AST (Investigations) | 1 (1)
Elevated blood pressure (Investigations) | 1 (1)
Elevated liver enzymes (Investigations) | 1 (1)
Fever (Investigations) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 1 (1)
Hypoalbuminemia (Metabolism and nutrition disorders) | 1 (1)
Hypocalcemia (Metabolism and nutrition disorders) | 1 (1)
Hypokalemia (Metabolism and nutrition disorders) | 2 (3)
Hypomagnesemia (Metabolism and nutrition disorders) | 1 (2)
Iron deficiency (Metabolism and nutrition disorders) | 1 (1)
Weight gain (Metabolism and nutrition disorders) | 1 (1)
Weight loss (Metabolism and nutrition disorders) | 7 (7)
Cramping - bilateral feet (Musculoskeletal and connective tissue disorders) | 1 (1)
Cramping - bilateral hands (Musculoskeletal and connective tissue disorders) | 1 (1)
Pain - abdominal (Musculoskeletal and connective tissue disorders) | 1 (1)
Pain - hip (Musculoskeletal and connective tissue disorders) | 4 (6)
Pain - jaw (Musculoskeletal and connective tissue disorders) | 1 (1)
Pain - lower back (Musculoskeletal and connective tissue disorders) | 2 (2)
Pain - muscles (Musculoskeletal and connective tissue disorders) | 1 (1)
Pain - right flank (Musculoskeletal and connective tissue disorders) | 1 (1)
Pain - shoulder (Musculoskeletal and connective tissue disorders) | 1 (1)
Pain - thighs (Musculoskeletal and connective tissue disorders) | 1 (1)
Weakness - legs (Musculoskeletal and connective tissue disorders) | 2 (2)
Disequilibrium (Nervous system disorders) | 1 (1)
Dizziness (Nervous system disorders) | 3 (3)
Headache (Nervous system disorders) | 3 (3)
Neuropathy (Nervous system disorders) | 1 (1)
Neuropathy - peripheral (Nervous system disorders) | 1 (1)
Neuropathy - sensory (Nervous system disorders) | 1 (1)
Pain - sinus (Nervous system disorders) | 1 (1)
Depression (Psychiatric disorders) | 1 (1)
Mental status change (Psychiatric disorders) | 1 (1)
Frequent urination (Renal and urinary disorders) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 6 (10)
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (2)
Pulmonary edema (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Alopecia (Skin and subcutaneous tissue disorders) | 4 (4)
Dry skin (Skin and subcutaneous tissue disorders) | 1 (1)
Erythema (Skin and subcutaneous tissue disorders) | 1 (1)
Erythema - face (Skin and subcutaneous tissue disorders) | 1 (1)
Erythema - feet (Skin and subcutaneous tissue disorders) | 1 (1)
Hand and foot syndrome (Skin and subcutaneous tissue disorders) | 1 (1)
Nail discoloration (Skin and subcutaneous tissue disorders) | 1 (1)
Numbness in face (Skin and subcutaneous tissue disorders) | 1 (1)
Onycholysis right thumbnail (Skin and subcutaneous tissue disorders) | 1 (1)
Pruritis / itching scalp (Skin and subcutaneous tissue disorders) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 4 (4)
Rash - back (Skin and subcutaneous tissue disorders) | 1 (1)
Rash - face (Skin and subcutaneous tissue disorders) | 1 (1)
Rash - generalized (Skin and subcutaneous tissue disorders) | 1 (1)
Rash - hand/foot/scalp (Skin and subcutaneous tissue disorders) | 1 (1)
Rash - mouth (Skin and subcutaneous tissue disorders) | 1 (1)
Rash - hand and foot (Skin and subcutaneous tissue disorders) | 1 (3)
Ruddy complexion (Skin and subcutaneous tissue disorders) | 1 (1)
Sensory neuropathy sensitivity - feet (Skin and subcutaneous tissue disorders) | 1 (1)
Skin irritation (Skin and subcutaneous tissue disorders) | 1 (1)
Tingling on scalp (Skin and subcutaneous tissue disorders) | 1 (1)
Stent placement (Surgical and medical procedures) | 1 (1)
Hypertension (Vascular disorders) | 4 (5)
Hypotension (Vascular disorders) | 2 (2)

LIMITATIONS AND CAVEATS:
Early termination, according to the stopping rule included in the protocol, leading to a small number of subjects analyzed

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Prior to publication or presentation of Sponsored Research results, Researcher agrees to provide Bayer with such presentation or manuscript at least 30 days prior to its submission for the sole purpose of allowing Bayer to redact confidential information and protect any existing or future patents. The Principal Investigator shall acknowledge Bayer contributions where appropriate.